CLINICAL TRIAL: NCT03084445
Title: Impact of Exposure to Environmental Pollutants on Birth Outcomes in an Israeli Cohort
Status: Active, not recruiting | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 12/12
Record Dates: First submitted 2014-02-06; First posted 2017-03-21 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Exposure to Environmental Pollution
Keywords: Brominated Flame Retardants (BFRs); Phthalates; pregnant women; newborn; Heavy Metals; Volatile Organic Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, red blood cells, urine, breast milk, meconium
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives and hypothesis The scale and diversity of chemicals in worldwide use today is vast. Many of these chemicals are released into the environment where they are found in air, water, soil, house dust, and in the food supply, resulting in exposure to humans. Characterizing the extent of exposure and the effects of exposure in vulnerable populations, such as pregnant women and children, is of the utmost importance as the chemical structure of many of these compounds resembles hormones such as estrogen, testosterone and thyroid hormone, affect neurodevelopment and other health effects. Here, we focus on few classes of compounds: heavy metals, volatile organic compounds (VOCs), brominated flame retardants (PBDEs) and phthalates. We will characterize the extent of exposure to pregnant women and their infants in Israel, where biomonitoring studies in the general population are scarce. We will also examine selected outcomes in pregnant women and their offspring in relation to these compounds, and to establish a biorepository for further studies.

Specific Aims:

1. To assess Heavy metals, VOCs, PBDEs and phthalates body burdens through measurement of these chemicals in maternal and paternal serum and urine, cord blood, breastmilk and neonatal meconium among several representative sub-populations.
2. To examine associations between exposure to heavy metals, VOCs, PBDEs and phthalates and (a) pregnancy complications, (b) anthropometrics at birth (i.e. birth weight adjusted for gestational age, ponderal index, head circumference adjusted for gestational age), and (c) cryptorchidism incidence, (d) maternal and infant thyroid function.
3. To establish a bio repository of these media for future studies and to establish follow up methods for this cohort to later assess development and growth in the infants, toddlers and children.

Patients and Methods:

Patients will be recruited from three delivery rooms in Israel: "Assaf Harofeh Medical Center" , "Lis (Sorasky) Medical Center" and "Rambam Medical Center", all together with around 21,000 births annually, representing all sub-populations in Israel. 500 mother-father-infant trios (for a total of 4500) will be recruited.

When arriving to the delivery room, after signing the informed consent, blood and urine will be withdrawn from the mothers and fathers for Heavy metals, VOCs, PBDEs and phthalates levels. At the same time thyroid function tests will also be taken from the mothers. After delivery, cord blood will be taken, as well as meconium from the neonate. Hair, nails and Breastmilk will also be collected. From the mothers The samples will be analyzed for heavy metals, VOCs, PBDEs and phthalates. During their stay at the hospital, mothers and fathers will fill out a standardized questionnaire regarding life style factors, background information, and exposure opportunities. Detailed information on family history, previous and present pregnancy, method of delivery, perinatal complications, and pregnancy outcome will be recorded from the medical files.

Expected contribution to environmental health in Israel:

This will be the first data on sub-populations exposure to Heavy metals, VOCs, PBDEs and phthalates in Israel. Neonatal meconium levels will provide important information on magnitude of exposure during the last months of pregnancy, and, thus, will provide insights into the bioaccumulative nature of these Heavy metals, VOCs, PBDEs and phthalates during early stages of human development, important data for future risk assessments. Our comprehensive approach will provide detailed information on the status of each subject. Such novel knowledge would also lead to the development of preventive and counseling strategies for men and women with high BFR and phthalates exposure in order to minimize the risks of adverse outcomes. Knowledge transfer strategies are essential in order that the general public, health professionals, scientists and policy/law regulators have the appropriate knowledge on which to base their understandings and recommendations for the future. In this way, the knowledge that is generated will facilitate the development of prevention strategies to minimize health risks of Israel population.

DETAILED DESCRIPTION:
Objectives and hypothesis The scale and diversity of chemicals in worldwide use today is vast, ranging from pharmaceuticals and food products, to plastics, gasoline, and semiconductor chips. Many of these chemicals are released into the environment where they are found in air, water, soil, in house dust, and in the food supply, resulting in exposure to humans. Characterizing the extent of exposure and the effects of exposure in vulnerable populations, such as pregnant women and children, is of the utmost importance as the chemical structure of many of these compounds resemble hormones such as estrogen, testosterone and thyroid hormone , affect neurodevelopment and other health effects. Here, we focus on few classes of compounds: heavy metals, volatile organic compounds (VOCs), brominated flame retardants (PBDEs) and phthalates., and will characterize the extent of exposure to pregnant women and their infants in Israel, where biomonitoring studies in the general population are scarce. We also propose to examine selected outcomes in pregnant women and their offspring in relation to these compounds, and to establish a biorepository for further studies.

BTEX (Benzene, Toluene, Ethylbenzene, Xylene):

Volatile organic compounds (VOCs) are compounds with low boiling points; VOC exposures originate from numerous natural and anthropogenic sources such as cleaning products, paints, solvents, personal care products, automotive exhaust, and tobacco smoke. Exposure to certain VOCs may increase the risk for birth defects, neurocognitive impairment, asthma, and cancer. The known VOC metabolites are acrolein, acrylamide, acrylonitrile, benzene, 1-bromopropane, 1,3-butadiene, carbon disulfide, crotonaldehyde, cyanide, N,N-dimethylformamide, ethylbenzene, ethylene oxide, propylene oxide, styrene, tetrachloroethylene, toluene, trichloroethylene, vinyl chloride, and xylene exposures. Benzene, toluene, ethylbenzene and xylene isomers (BTEX), aromatic hydrocarbons, are part of VOC metabolites that play a major role in industries and air pollution 1.

Prena¬tal exposure to air pollution (contains BTEX) might be associated with adverse pregnancy outcomes, including intrauterine growth restriction (IUGR), low birth weight (LBW), preterm birth (PTB), and intrauter¬ine mortality. Exposure to BTEX chemicals has been associated with negative impacts on sperm quantity and quality. Benzene and toluene exposure have been associated with abnormal menstrual cycle. Direct adverse effects of BTEX chemicals have been observed on ovarian cell apoptosis, proliferation, and hormone release in animal ovarian cells. Exposures to benzene and toluene, commonly used and produced by unconventional oil and gas (UOG) operations, have been associated with increased risks for miscarriage 2.

Xylene is an environmental pollutant. It is also used in dyes, paints, polishes, medical technology and different industries as a solvent. Human life is surrounded by a wide range of VOCs, including xylene causing harmful health effects xylene exposure occurs through breath, eye, oral, and dermal route. Xylene is mainly metabolized in the liver via oxidation of methyl groups, followed by conjugation with glycine to yield hippuric acid, which is excreted through urine. High amount and dose of xylene may harm the liver. Prolonged exposure to xylene may cause a multiorgan damages such as: toxicity to nervous, reproductive, immune, hepatic and respiratory systems. Furthermore, xylene reduces reproductive hormones in women and cause male infertility. Studies have reported the subsequent effects in experimental animals: deformities in fetus skeletal, increased interruption in bone formation, redness and blood in fetus organs, and reduced fetus weight3.

Benzene is known as one of the predominant air pollutants in the environment. Chronic exposure to benzene is known to cause oxidative stress, DNA damage, aplastic anemia and increased risk of acute myelogenous leukemia in humans. The mechanism is through crucial toxic metabolism, reactive metabolites and probably epigenetic changes. Common exposures to benzene are tobacco smoke, automobile service stations, exhaust from motor vehicles, and industrial emissions. Chromosomal abnormalities in sperm have also been reported with benzene exposure4 [4],

Ethylbenzene originates from tobacco smoke, burning fossil fuels, industries using ethylbenzene, carpet glues, varnishes and paints. The hazards of ethylbenzene include acute toxicity, mutagenicity, systemic toxicity, developmental and reproductive toxicity, immunotoxicity, metabolism and pharmacokinetics, carcinogenicity, neurotoxicity, and developmental neurotoxicity. At doses that produced maternal effects (> 1000 ppm) in animals, ethylbenzene was fetotoxic causing decreased fetal body weight (bwt) and increased skeletal variations5.

Exposure to toluene is from, industrial paints and paint thinner, tobacco smoke, and fossil fuels6. Toluene has intoxicating and rewarding effects in the brain. Acute exposure to inhalants has dose dependent, reversible effects like depressed central nervous system (CNS). High concentrations can cause sedation and anesthesia, while higher concentration can result in coma or death by respiratory depression. At delivery, toluene-exposed infants were characteristically premature and/or delayed in growth as. Additionally, as the children grow, a number of developmental delays and impairments become evident (e.g., language impairments, growth retardation, hyperactivity, cerebellar dysfunction)7.

Trichloroethylene (TCE) and perchloroethylene (PCE) are part of the VOCs and the air pollution. It is known that the risk of epilepsy and certain types of cancer such as cervical cancer may be increased among adults who were exposed to PCE-contaminated drinking water. Exposure during gestation and early childhood and exposure to a major metabolite of TCE, TCAA (trichloroacetic acid)administered in drinking water, resulted in increased numbers of implantation and resorption sites, and selective cardiac teratogenicity8,9.

Heavy metal elements:

Metal intake can be via air, water and food. Air pollution exposure includes inhalation or ingestion of ultrafine particulate matter, also called nanoparticles. Epidemiological studies have consistently found an association between small increases in urban particulates and health effects, including increased morbidity and mortality in people with respiratory and cardiac disease. All metals in excess can cause disease. Long term exposure to metal is a cause of increased metal accumulation in a variety of body tissue. Some metals are more toxic than others10.

The prevalent elements that found in soil in Haifa bay:

* Nickel (Ni) - Nickel sensitivities are the most common harmful health effect in humans. People working in nickel refineries or nickel-processing plants are more affected with chronic bronchitis, asthma and reduced lung function then the general population.
* Lead (Pb) - neurological ailments and learning impairments can inactive enzymes, thus affecting red blood cell production, amino acid function and number of biochemical systems in the body. Lead exposure is associated with an increased risk of miscarriage and stillbirth potentially due to placental rupture.
* Chromium (Cr) - is found in all phases of the environment including air, water, and soil, and its many chemical forms are pollutants with serious implication to the environment and human health. Hexavalent chromium (Cr6) occurs in the environment from the erosion of natural chromium deposits, but is also a product of industrial processes. There are demonstrated instances of Cr6 being released into the environment by leakage, poor storage, or inadequate industrial waste disposal practices.
* Mercury (Hg) - affects central nervous function. A source of it is an exposure to breathing air from spills, incinerators and industries burning mercury containing fuels. Mercury, at high levels, may damage the brain, kidneys, and the developing fetus. Short-term exposure to high levels of metallic mercury vapors may cause lung damage, nausea, vomiting, diarrhea, increases in blood pressure or heart rate, skin rashes, and eye irritation11.
* Cadmium- elevated cadmium exposure during pregnancy may be inversely associated with children's cognitive function measured at pre-school age. Exposure to cadmium has been shown to result in miscarriage and stillbirths in exposed mothers, potentially through decreased levels of antioxidants or enhanced lipid peroxidation resulting in oxidative stress12.
* Mangenase (Mn) - is used in steel production to improve hardness, stiffness, and strength. It may be used as an additive in gasoline to improve the octane rating of the gas. Exposure to high level of manganese in air can cause lung irritation and reproductive effects.13 The central nervous system is a common target organ for many environmental metals. The adverse effects of heavy metal exposure in the prenatal and early childhood periods are of increasing concern in terms of high exposure on a body weight basis, immature metabolic pathways, delicate developmental processes, and life course effects. Prenatal exposure to lead and mercury has been related to congenital anomalies and impaired neurodevelopment. Metals may interact to cause synergistic or antagonistic effects on neurodevelopment that are different from the main effects of exposure to each metal alone. Metals exposure during prenatal and childhood may affect the neurodevelopment/cognitive and behavior14.

If more risk factors such as genetic, ethnic and environmental exposure coincide, disease development is more likely to progress. Exposure to heavy metals during pregnancy is associated with increased risks of miscarriage and/or stillbirths.

Heavy metals may be routinely mobilized during hydraulic fracturing operations and have been shown to contaminate surface and ground water in some cases (e.g., lead), they are also inadvertent contaminants in fracturing fluids.

Brominated Flame Retardants Brominated Flame Retardants (BFRs) constitute a group of chemical substances that are used worldwide to reduce fire-related injury and property damage. They are found in polymers (polystyrene foams, high impact polystyrene, epoxy resins) that are incorporated into a wide variety of consumer products (textiles, foam furniture, insulating foams, electrical equipment, kitchen appliances, televisions and computers). In 2000, it was estimated that >200,000 metric tons of BFRs were produced annually. There are currently five major BFRs: three commercial mixtures of polybrominated diphenyl ethers (penta-, octa- and deca-BDEs), hexabromocyclododecane (HBCD) and tetrabromobisphenol A (TBBPA) routinely present in a broad variety of consumer goods. Because BFRs leach out of manufactured products and these products are dumped in the environment, we are exposed to BFRs from a wide variety of sources.

The concentration of BFRs in the environment, has increased dramatically over the past two decades while, thanks to international regulatory policies, that of other known toxicants (DDT, lead, PCBs) has declined.

Exposure through contaminated food, particularly meat and dairy products, is believed to be the major contributor to BFR exposure in humans.

There are reports that newborns and young infants have higher serum concentrations than older children and adults, since it is generally believed that infants are more vulnerable to toxicological insults. Scientists in the USA have reported that the median levels of BDEs in human breast milk increased almost 10-fold from the 90's to the early 2000's. The in-utero period is a critical period for exposure; however, there is a scarcity of information with respect to BFR exposure during the earliest stages of human development. A study monitoring tetra- to octa-BDE levels in early to mid-gestation human fetal liver and placenta from 1998-2006, demonstrated not only that these toxicants cross the placenta from as early as nine weeks fetal age but also that the 2006 fetal tissue levels are >5-fold higher than they were nine years previously. Thus, fetal BFR exposure is also on the rise.

Although the BFR burden in humans is increasing and exposures occur from an early stage in development, the consequences are relatively unexplored. Three clinical studies have been published to date on the potential effects of in-utero BFR exposure and fetal outcome. Elevated levels of BFRs in breast milk correlated significantly with lower newborn birth weight, birth length, head size, chest circumference and body mass index. Significant associations between maternal serum BFR levels at 35 weeks gestation and the levels of several sex hormones (testosterone, estradiol, LH, SHBG) in 3 month old female and male offspring were reported. In addition, Main and colleagues have found significantly higher BFR levels in the breast milk of mothers whose newborn sons had cryptorchidism. If left untreated, cryptorchidism can lead to serious reproduction-related problems: low sperm counts and infertility as well as a 2- to 8-fold increase in the risk of testicular cancer. These data suggest that BFRs are impacting early stages of human development and that at least one outcome is abnormal reproductive systems. This is a serious issue: not only is an individual's health potentially affected but so is that of future generations.

Phthalates Phthalates are a class of high production volume chemicals used in a wide variety of consumer products. They are commonly used as plasticizers to increase flexibility and durability. They are also used to hold fragrances, and as propellants. Global production of phthalates has increased dramatically since World War II and is currently estimated to exceed 3.5 million metric tons/year. DEHP constitutes roughly 50% of the market share, but uses of DBP and BBzP are also large (> 100,000 metric tons/year each). The widespread use has resulted in ubiquitous contamination, including of the indoor environment, with exposures higher in industrialized than in developing nations. Table 1 below shows sources of exposure of the phthalate diesters that will be evaluated in the proposed study.

Some recent studies, find prenatal exposure to phthalates to be associated with reductions in fetal growth, shorter pregnancy duration, perturbed thyroid function, and both cognitive and behavioral deficits in children. More data are clearly required to fully characterize the health effects in vulnerable populations of pregnant women and children.

Specific Aims:

1. To assess Heavy metals, VOCs, PBDEs and phthalates body burdens through measurement of these chemicals in maternal and paternal serum and urine, cord blood, breastmilk and neonatal meconium among several representative sub-populations.
2. To examine associations between exposure to heavy metals, VOCs, PBDEs and phthalates and (a) pregnancy complications, (b) anthropometrics at birth (i.e. birth weight adjusted for gestational age, ponderal index, head circumference adjusted for gestational age), and (c) cryptorchidism incidence, (d) maternal and infant thyroid function.
3. To establish a bio repository of these media for future studies and to establish follow up methods for this cohort to later assess development and growth in the infants, toddlers and children.

Patients and Methods:

Patients will be recruited from three delivery rooms in Israel: "Assaf Harofeh Medical Center" , "Lis (Sorasky) Medical Center" and "Rambam Medical Center", all together with around 21,000 births annually, representing all sub-populations in Israel. 500 mother-father-infant trios (for a total of 4500) will be recruited.

When arriving to the delivery room, after signing the informed consent, blood and urine will be withdrawn from the mothers and fathers for Heavy metals, VOCs, PBDEs and phthalates levels. At the same time thyroid function tests will also be taken from the mothers. After delivery, cord blood will be taken, as well as meconium from the neonate. Hair, nails and Breastmilk will also be collected. From the mothers The samples will be analyzed for heavy metals, VOCs, PBDEs and phthalates. During their stay at the hospital, mothers and fathers will fill out a standardized questionnaire regarding life style factors, background information, and exposure opportunities. Detailed information on family history, previous and present pregnancy, method of delivery, perinatal complications, and pregnancy outcome will be recorded from the medical files.

Feasibility of the research:

Delivery, maternal and neonatal departments in all medical centers have a large number of deliveries annually. The population admitted to these centers is representative of the population in Israel. Since blood work is part of the admission to the delivery room, and since the neonates will not have an invasive procedure (meconium), we expect many couples to participate in this innovative study. Our comprehensive approach, using a combination of a standardized questionnaire, maternal and paternal serum, cord blood, urine, breastmilk and meconium analysis of the chemicals, will provide a detailed definition of the body burden status of each subject. We have the means and the desire to facilitate knowledge exchange between basic and clinical scientists, between those who generate knowledge and those who use it in developing policies and regulations, as well as among scientists, health professionals and the general public.

Expected contribution to environmental health in Israel:

These will be the first data on sub-populations exposure to Heavy metals, VOCs, PBDEs and phthalatesin Israel. Neonatal meconium levels will provide important information on magnitude of exposure during the last months of pregnancy, and, thus, will provide insights into the bioaccumulative nature of these Heavy metals, VOCs, PBDEs and phthalatesduring early stages of human development, important data for future risk assessments. Our comprehensive approach will provide detailed information on the status of each subject. Such novel knowledge would also lead to the development of preventive and counseling strategies for men and women with high BFR and phthalate exposure in order to minimize the risks of adverse outcomes. Knowledge transfer strategies are essential in order that the general public, health professionals, scientists and policy/law regulators have the appropriate knowledge on which to base their understandings and recommendations for the future. In this way, the knowledge that is generated will facilitate the development of prevention strategies to minimize health risks of Israel population.

ELIGIBILITY:
Inclusion Criteria:

* Israeli Arabs, Jews from Russia, Jews from Ethiopia, Jews with an Ashkenazic background and Jews with a Sephardic background

Exclusion Criteria:

* refuse to take part in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women and their partners attenting delivery room
Sampling Method: Non-Probability Sample
Enrollment: 2394 (Actual)
Dates: Start 2013-09; Primary Completion 2020-06 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring envinromental polutants, including heavy metals, VOCs, PBDEs and phthalates levels in collected samples | 48 months after end of specimens collection
  assessment of BFRs and phthalates body burdens through measurement of these chemicals in maternal and paternal serum and urine, cord blood, breastmilk and neonatal meconium among several representative sub-populations

SECONDARY OUTCOMES:
associations between exposure to nvinromental polutants, including heavy metals, VOCs, PBDEs and phthalates and few maternal and infant pregnancy and birth parameters and endocrine functions | 48 months after end of specimens collection
  To examine associations between exposure to PBDEs and phthalates and (a) pregnancy complications, (b) anthropometrics at birth (i.e. birth weight adjusted for gestational age, ponderal index, head circumference adjusted for gestational age), and (c) cryptorchidism incidence, (d) maternal and infant thyroid function

OTHER OUTCOMES:
To establish a bio repository of these media for future studies | 15 years after end of specimens collection
  To establish a bio repository of these media for future studies and to establish follow up methods for this cohort to later assess development and growth in the infants, toddlers and children

CONTACTS AND LOCATIONS:
Overall Officials: Mati Berkovitch, Prof., Principal Investigator — Assaf-Harofeh Medical Center
Locations (3):
- Israel (3):
  - Rambam Medical Center, Haifa
  - Lis Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin